CLINICAL TRIAL: NCT05368220
Title: TRANSLATE - Translating Genetic Knowledge Into Clinical Care in Non-Autoimmune Diabetes
Brief Title: Translating Genetic Knowledge Into Clinical Care in Non-Autoimmune Diabetes
Acronym: TRANSLATE
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other); BGI Europe (Unknown); Intomics A/S (Unknown); Rigshospitalet, Denmark (Other); Danish National Genome Center (Unknown); Nordsjaellands Hospital (Other); Herlev Hospital (Other); Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Torben Hansen, Professor, University of Copenhagen
Other Study IDs: 9090-00078B
Record Dates: First submitted 2022-05-02; First posted 2022-05-10 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes, Gestational
Keywords: Precision medicine; Personalized medicine; Genetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes, Gestational | interventions — Whole Genome Sequencing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Two 10ml EDTA blood tubes are collected, from which buffy coat is isolated and DNA is extracted for whole genome sequencing and quality control. Samples are stored for up to two years in order to repeat the analysis before being destroyed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with non-autoimmune diabetes (type 2 diabetes): Any case of non-T1D defined as:
  * Debut >30 years of age OR
  * Debut <30 years of age AND negative autoantibodies
  treated at Steno Diabetes Center Copenhagen
  Interventions: Other: Whole genome sequencing
- Patients with gestational diabetes: Any case of diabetes diagnosed in pregnancy treated at the following obstetric clinics in the Capital Region in Denmark:
  Rigshospitalet, Nordsjællands Hospital, Herlev Hospital, Hvidovre Hospital
  Interventions: Other: Whole genome sequencing

INTERVENTIONS:
Other: Whole genome sequencing — Each participant will have WGS performed in order to report on clinically actionable genetic variation in diabetes.
  Other Names: WGS

SUMMARY:
The aim of TRANSLATE is to implement genetic information directly into patient care to improve diagnosis and treatment of non-autoimmune diabetes. This project is the first large-scale implementation of systematic genetic testing within a common, non-communicable, chronic disease in Denmark, and will spearhead efforts to advance personalized medicine in Denmark.

The project will contribute to establishing technology, workflow, and evidence on how to implement and communicate actionable genetic information to clinicians and patients in a generalized format. These developments are pivotal for personalized medicine to reach broader clinical application.

DETAILED DESCRIPTION:
The TRANSLATE project is an integrative project with multifaceted goals, that can be broken down into two main columns. The foundation for both columns is the WGS analysis in a clinical diagnostic setting in order to guide patient treatment. Patients are not randomized and the inclusion and exclusion criteria are deliberately broad and minimal, respectively.

The first column is the clinical development project, which seeks to complete a novel diagnostic process. This column will develop new pipelines and uncover barriers and challenges associated with gene-based precision medicine to facilitate sustainable implementation of gene-based precision medicine beyond the TRANSLATE project.

During the project, we wish to focus on potential barriers against a broad application of gene-based precision medicine in a common disease. These may include:

* Challenges pertaining to the selection of variants that are deemed clinically actionable, automation of genetic interpretation/translation, and the feasibility of large-scale precision medicine implementation
* Ethical concerns of patients, clinicians, and other technicians with regard to the application and utility of genetic information
* Validity and limitations of current computational pipelines for variant calling including the calling of structural variants and aggregate genetic tools
* Challenges regarding the interoperability of IT systems and databases nationally in Denmark, specifically how central databases can be linked to clinical end-users
* How implementation of genetic analyses affects clinical decision-making and/or clinical trajectories, both qualitatively and quantitatively

The second column is a register-based research project in which we will utilize data from the patients to advance gene-based precision medicine. In this column we will both address how to establish comprehensive research infrastructure, as well as answer specific research questions. We will address how to combine and harmonize genetic data with other Danish registry sources. We will use the newly established methodologies to focus on the following research areas with respect to patient stratification, clinical trajectories, complication development, and other clinically relevant outcomes:

* Polygenic risk scores
* Machine learning algorithms
* Combined polygenic and monogenic traits
* Non-coding variation
* Structural variation, specifically exon deletions and duplications, which have previously been shown as a cause of monogenic diabetes

ELIGIBILITY:
Inclusion Criteria:

* Any case of non-T1D defined as debut >30 years of age, OR debut <30 years of age AND negative autoantibodies
* Any case of diabetes diagnosed in pregnancy (obstetric departments)

Exclusion Criteria:

* Age <18 years
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in the target groups with non-autoimmune/non-T1D attending SDCC or pregnant women with gestational diabetes attending one of the obstetric clinics in the project will be offered a genetic test.
Sampling Method: Non-Probability Sample
Enrollment: 6500 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Selection of clinically actionable genetic variation in diabetes | Until final patient inclusion (May 2025) + 2 years (May 2027)
  Using mixed methods such as gene burden investigations, workgroups, interviews, etc. challenges related to the selection of clinically actionable genetic variants and automation of interpretation/translation will be delineated.
Ethical concerns regarding the application and utility of genetic information | Until final patient inclusion (May 2025) + 2 years (May 2027)
  The project will address how patients, clinicians, technicians etc. shape their understanding of the utility and challenges associated with gene-based precision medicine using ethnographic methods such as field observations and semi-structured interviews.
Validity and limitations of current computational pipelines | Until final patient inclusion (May 2025) + 2 years (May 2027)
  By comparing computational and analytical methods, the project will investigate the validity and limitations of different computational pipelines. This includes handling of single nucleotide variants, as well as structural variation.
Interoperability of IT systems and databases | Until final patient inclusion (May 2025) + 2 years (May 2027)
  The project will address the flow of data to and from clinical end-users, through centralized databases, both with respect to how the data flow is perceived by users and potential challenges, and how interoperability can be improved to enhance clinical utility. The project will also address how to harmonize data from different sources.
Impact on clinical decision-making and clinical trajectories | Until final patient inclusion (May 2025) + 2 years (May 2027)
  Using mixed methods such as mapping of clinical trajectories through clinical registries and qualitative methods such as interviews, workgroups, etc., the project will investigate how implementation of gene-based precision diabetes impacts clinical decision making.

CONTACTS AND LOCATIONS:
Overall Officials: Torben Hansen, PhD, Principal Investigator — University of Copenhagen
Locations (5):
- Denmark (5):
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - Steno Diabetes Center Copenhagen, Herlev
  - Hillerød Hospital, Hillerød
  - Hvidovre Hospital, Hvidovre

IPD SHARING:
Plan to Share IPD: No
Data will be reported to Danish National Genome Center after completion.

REFERENCES:
- See also: Study website — http://translate.ku.dk